CLINICAL TRIAL: NCT00811941
Title: A 52-week, Randomised, Double-blind, Placebo-controlled, Parallel-group, Safety, Tolerability and Efficacy Study of Nalmefene, as Needed Use, in Patients With Alcohol Dependence
Brief Title: Safety and Efficacy of Nalmefene in Patients With Alcohol Dependence
Acronym: SENSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12013A; 2007-002315-92 (EudraCT Number)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-07

CONDITIONS: Alcohol Dependence
Keywords: Pharmacologic Actions; Alcohol-Related Disorders; Alcoholism; Mental Disorders; Central Nervous System Agents
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Mental Disorders | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Nalmefene (Experimental)
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Placebo — as-needed use, tablets, orally, 52 weeks
  Arms: Placebo
Drug: Nalmefene — 18.06 mg as-needed use, tablets, orally, 52 weeks. 18.06 mg nalmefene equals 20 mg nalmefene hydrochloride.
  Other Names: Selincro™
  Arms: Nalmefene

SUMMARY:
The purpose of the study is long-term safety, tolerability and efficacy of nalmefene in patients with alcohol dependence.

DETAILED DESCRIPTION:
Alcohol dependence is a maladaptive pattern of alcohol use, leading to clinically significant impairment or distress, as manifested by at least three of a number of criteria such as tolerance, withdrawal symptoms, frequent use of alcohol in larger amounts or over longer periods than was intended, and others. Excessive intake of alcohol reduces the life span by a decade, and alcohol drinking is strongly related to mortality from liver cirrhosis, chronic pancreatitis, certain cancers, hypertension, accidents and violence. This study is planned to evaluate the long-term safety and tolerability as well as to evaluate the efficacy of as needed use of 18.06 mg nalmefene in patients with alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

In- and outpatients who:

* had a primary diagnosis of alcohol dependence according to Diagnostic and Statistical Manual of Mental Disorders - text revision (DSM-IV-TR) criteria
* had had ≥6 Heavy Drinking Days (HDDs) in the 4 weeks preceding the Screening Visit

Exclusion Criteria:

The patient:

* had a severe psychiatric disorder or an antisocial personality disorder
* had risk of suicide evaluated by the suicidality module of the Mini-International Neuropsychiatric Interview (MINI)
* had a history of delirium tremens or alcohol withdrawal seizures
* reported current or recent (within 3 months preceding screening) treatment with disulfiram, acamprosate, topiramate, naltrexone or carbimide, or with any opioid antagonists
* was pregnant or breast-feeding

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2009-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (60):
- Czechia (5):
  - CZ007, Litoměřice
  - CZ006, Lnáře
  - CZ005, Prague
  - CZ004, Prague
  - CZ001, Ústí nad Labem
- Estonia (5):
  - EE002, Pärnu
  - EE004, Tallinn
  - EE005, Tallinn
  - EE003, Vorumaa
  - EE001, Võru
- Hungary (2):
  - HU004, Budapest
  - HU002, Budapest
- Latvia (4):
  - LV003, Daugavpils
  - LV002, Jelgava
  - LV001, Riga
  - LV004, Sigulda
- Lithuania (2):
  - LT002, Kaunas
  - LT003, Kaunas
- Poland (15):
  - PL015, Bełchatów
  - PL008, Bydgoszcz
  - PL006, Gdansk
  - PL011, Krakow
  - PL002, Leszno
  - PL010, Lodz
  - PL014, Lodz
  - PL004, Lublin
  - PL005, Lublin
  - PL013, Piekary Śląskie
  - PL003, Skorzewo
  - PL007, Starogard Gdański
  - PL012, Swicie n/Wisla
  - PL009, Szczecin
  - PL001, Torun
- Russia (8):
  - RU013, Rostov-on-Don
  - RU002, Saint Petersburg
  - RU005, Saint Petersburg
  - RU006, Saint Petersburg
  - RU001, Saint Petersburg
  - RU012, Saint Petersburg
  - RU003, Saint Petersburg
  - RU004, Voronezh
- Slovakia (4):
  - SK001, Banska Bysterica
  - SK002, Krupina
  - SK004, Nitra
  - SK005, Rimavská Sobota
- Ukraine (10):
  - UA001, Chernihiv
  - UA008, Dnipropetrovsk
  - UA003, Donetsk
  - UA004, Hlevakha
  - UA007, Kharkiv
  - UA009, Kherson
  - UA002, Kyiv
  - UA005, Odesa
  - UA006, Simferopol
  - UA010, Ternopil
- United Kingdom (5):
  - GB007, Birmingham
  - GB006, Glasgow
  - GB009, London
  - GB008, Manchester
  - GB005, Reading

REFERENCES:
- [Derived] Laramee P, Brodtkorb TH, Rahhali N, Knight C, Barbosa C, Francois C, Toumi M, Daeppen JB, Rehm J. The cost-effectiveness and public health benefit of nalmefene added to psychosocial support for the reduction of alcohol consumption in alcohol-dependent patients with high/very high drinking risk levels: a Markov model. BMJ Open. 2014 Sep 16;4(9):e005376. doi: 10.1136/bmjopen-2014-005376. PMID 25227627

RESULTS

PARTICIPANT FLOW:
Groups:
- Nalmefene 18.06 mg: as-needed use, tablets, orally, 52 weeks
Period: All Randomised Patients
Arm/Group | Placebo | Nalmefene 18.06 mg
Started | 166 | 509
Completed | 164 | 501
Not Completed | 2 | 8
Not completed — Did not receive placebo/nalmefene | 2 | 8
Period: All Treated Patients
Arm/Group | Placebo | Nalmefene 18.06 mg
Started | 164 | 501
Completed | 112 (Patients who had the final visit of the study protocol) | 310 (Patients who had the final visit of the study protocol)
Not Completed | 52 | 191
Not completed — Adverse Event | 2 | 43
Not completed — Lack of Efficacy | 2 | 3
Not completed — Non-compliance | 1 | 8
Not completed — Protocol Violation | 5 | 17
Not completed — Withdrawal by Subject | 35 | 94
Not completed — Lost to Follow-up | 3 | 12
Not completed — Other Reason | 4 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nalmefene 18.06 mg | Total
Number analyzed (Participants) | 166 | 509 | 675
Age Continuous [Mean (Standard Deviation); unit: years] — All-patients-randomised set (APRS).
  years | 44.3 (12.0) | 44.3 (11.2) | 44.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — APRS.
  Participants
    Female | 39 | 116 | 155
    Male | 127 | 393 | 520
Previously Treated for Alcohol Dependence [Number; unit: participants] — APRS.
  participants
    NO | 105 | 338 | 443
    YES | 61 | 171 | 232
Previously Treated for Alcohol Withdrawal Symptoms [Number; unit: participants] — APRS.
  participants
    NO | 118 | 372 | 490
    YES | 48 | 137 | 185
Total Monthly Heavy Drinking Days (HDD) [Mean (Standard Deviation); unit: days] — APRS.
  Based on Timeline Followback (TLFB) data from the month preceding the screening visit.
  days | 13.69 (6.03) | 14.08 (6.22) | 13.98 (6.17)
Total Alcohol Consumption (TAC) g Alcohol/Day [Mean (Standard Deviation); unit: g] — APRS.
  Based on TLFB data from the month preceding the screening visit.
  g | 68.00 (40.62) | 68.64 (39.98) | 68.49 (40.11)
Drinking Risk Level (DRL) [Number; unit: participants] — APRS.
  participants
    UNKNOWN | 0 | 1 | 1
    LOW | 26 | 79 | 105
    MEDIUM | 49 | 167 | 216
    HIGH | 59 | 148 | 207
    VERY HIGH | 32 | 114 | 146
Clinical Global Impression - Severity of Illness (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — APRS.
  The Clinical Global Impression - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 3.88 (1.03) | 3.95 (1.12) | 3.94 (1.09)
Gamma-glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: international units per liter (IU/L)] — APRS.
  international units per liter (IU/L) | 71.03 (116.25) | 68.82 (109.87) | 69.36 (111.39)
Alanine Aminotransferase (ALAT) [Mean (Standard Deviation); unit: IU/L] — APRS.
  IU/L | 31.46 (20.20) | 33.87 (22.61) | 33.28 (22.05)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: Overview of AEs
Time Frame: Serious Adverse Events: 52 weeks and a safety follow-up (visit/telephone call) scheduled for 4 weeks after completion of the study or after withdrawal from the study. Other Adverse Events: 52 weeks.
Population: All-patients-treated set (APTS) - all patients in the APRS excluding those with no recorded investigational medicinal product (IMP) intake and all IMP returned
Measure: Number; unit: participants
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 164 | 501
participants
  Patients with AEs | 103 | 377
  Patients with Serious AEs (SAEs) | 8 | 35
  Patients with AEs Leading to Withdrawal | 5 | 57

2. Primary Outcome: Percentage of Patients Who Withdrew Due to Intolerance to Treatment
Time Frame: Baseline to Week 52
Population: All-patients-treated Set (APTS)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 164 | 501
percentage of participants | 1.2 | 8.6

3. Primary Outcome: Change From Baseline in the Monthly Number of Heavy Drinking Days (HDDs)
Description: Number of HDDs over a month (28 days), where one HDD was defined as a day with alcohol consumption ≥60 grams (g) for men and ≥40 g for women.
Time Frame: Baseline and Month 6
Population: Full-analysis set (FAS) - all patients in the APTS who had at least one valid post-baseline assessment in the main treatment period of both co-primary efficacy variables (HDD and TAC) and had an average alcohol consumption at medium Drinking Risk Level (DRL) or above according to WHO criteria at Baseline.
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 110 | 320
days | -8.92 (0.56) | -9.80 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; The primary hypothesis concerned the treatment effect at Month 6. Null hypothesis of no difference in treatment effect was tested against the alternative hypothesis that there was a difference in treatment effect. MMRM model with the Baseline score as a covariate; site, sex, time in months (Month 1-13); and treatment as fixed effects. The Baseline score-by-time and treatment-by-time interactions were also included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.160, Adjusted change from Baseline to Month 6; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-2.10 to 0.35], Standard Error of Mean 0.62 — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 110 participants in the placebo group and 320 participants in the nalmefene group

4. Primary Outcome: Change From Baseline in the Monthly Total Alcohol Consumption (TAC)
Description: TAC was defined as mean daily alcohol consumption in g/day over a month (28 days).
Time Frame: Baseline and Month 6
Population: FAS
Measure: Mean (Standard Error); unit: g
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 110 | 320
g | -45.58 (2.61) | -49.05 (1.64)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; The primary hypothesis concerned the treatment effect at Month 6. The null hypothesis of no difference in treatment effect was tested against the alternative hypothesis that there was a difference in treatment effect. MMRM model with the Baseline score as a covariate; site, sex, time in months (Month 1-13); and treatment as fixed effects. The Baseline score-by-time and treatment-by-time interactions were also included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.232, Adjusted change from Baseline to Month 6; Mean Difference (Final Values) = -3.47, 95% CI 2-sided [-9.17 to 2.23], Standard Error of Mean 2.90 — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Drinking Risk Level (RSDRL) Response
Description: RSDRL response was defined as a downward shift from baseline in Drinking Risk Level (DRL); for patients at very high risk at Baseline: a shift to medium risk or below, and for patients at high or medium risk at Baseline: a shift to low risk or below.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 137 | 415
percentage of participants | 63.5 | 62.2
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; The analysis of RSDRL used a logistic regression (LREG) model, with country, sex, Baseline DRL, and treatment as fixed effects, and missing values were imputed using individual-patient predicted values of TAC derived from the MMRM model; Test type: Superiority or Other; p = 0.689, Adjusted Odds Ratio (OR) response; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.59 to 1.41]

6. Secondary Outcome: Change From Baseline in Clinical Status Using CGI-S
Description: The Clinical Global Impression - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline and Week 24
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 104 | 306
units on a scale | -0.75 (0.08) | -0.94 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; MMRM model with the Baseline score as a covariate, and site, sex, time in weeks, and treatment as fixed effects. The Baseline score-by-time and treatment-by-time interactions were also included in the model; an unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.046, Adjusted change from Baseline to Week 24; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.37 to -0.00], Standard Error of Mean 0.09 — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 104 participants in the placebo group and 306 participants in the nalmefene group

7. Secondary Outcome: Change in Clinical Status Using the CGI-I
Description: The Clinical Global Impression - Global Improvement (CGI-I) provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7- point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 24
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 104 | 306
units on a scale | 2.68 (0.10) | 2.54 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; MMRM model with the Baseline CGI-S score as a covariate, and site, sex, time in weeks, and treatment as fixed effects. The Baseline CGI-S score-by-time and treatment by- time interactions were also included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.217, Adjusted change from Baseline to Week 24; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.36 to 0.08], Standard Error of Mean 0.11 — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Liver Function Test Gamma-glutamyl Transferase (GGT)
Description: GGT values
Time Frame: Week 24
Population: FAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 108 | 319
IU/L | 34.5 (63.5) | 32.2 (71.1)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; Log-transformed GGT values were analysed using an MMRM model with the logtransformed Baseline value as a covariate, and site, sex, time in weeks, and treatment as fixed effects. Log-transformed Baseline value-by-time interaction and treatment-by-time interaction were included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.273, Adjusted values; Ratio to placebo = 0.93, 95% CI 2-sided [0.83 to 1.05] — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 108 participants in the placebo group and 319 participants in the nalmefene group

9. Secondary Outcome: Liver Function Test Alanine Aminotransferase (ALAT)
Description: ALAT values
Time Frame: Week 24
Population: FAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 108 | 318
IU/L | 25.8 (52.4) | 25.6 (56.7)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; Log-transformed ALAT values were analysed using an MMRM model with the logtransformed Baseline value as a covariate, and site, sex, time in weeks, and treatment as fixed effects. Log-transformed Baseline value-by-time and treatment-by-time interactions were included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.916, Adjusted values; Ratio to placebo = 0.99, 95% CI 2-sided [0.90 to 1.10] — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 108 participants in the placebo group and 318 participants in the nalmefene group

10. Secondary Outcome: Change From Baseline in the Monthly Number of Heavy Drinking Days (HDDs)
Description: Number of HDDs over a month (28 days), where one HDD was defined as a day with alcohol consumption ≥60 g for men and ≥40 g for women.
Time Frame: Baseline and Month 13
Population: FAS
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 97 | 258
days | -8.96 (0.58) | -10.53 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; MMRM model with the Baseline score as a covariate; site, sex, time in months (Month 1-13); and treatment as fixed effects. The Baseline score-by-time and treatment-by-time interactions were also included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.017, Adjusted change from Baseline - Month 13; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-2.85 to -0.29], Standard Error of Mean 0.65 — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 97 participants in the placebo group and 258 participants in the nalmefene group

11. Secondary Outcome: Change From Baseline in the Monthly Total Alcohol Consumption (TAC)
Description: TAC was defined as mean daily alcohol consumption in g/day over a month (28 days).
Time Frame: Baseline and Month 13
Population: FAS
Measure: Mean (Standard Error); unit: g
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 97 | 258
g | -46.33 (2.73) | -52.80 (1.76)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.036, Adjusted change from Baseline - Month 13; Mean Difference (Final Values) = -6.47, 95% CI 2-sided [-12.53 to -0.42], Standard Error of Mean 3.07 — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Drinking Risk Level (RSDRL) Response
Description: as for outcome 5
Time Frame: Month 13
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 137 | 415
percentage of participants | 54.0 | 54.5
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.976, Adjusted Odds Ratio (OR) response; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.67 to 1.52]

13. Secondary Outcome: Change From Baseline in Clinical Status Using CGI-S
Description: as for outcome 6
Time Frame: Baseline and Week 52
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 95 | 258
units on a scale | -1.08 (0.10) | -1.30 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.056, Adjusted change from Baseline to Week 52; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.44 to 0.01], Standard Error of Mean 0.11 — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 95 participants in the placebo group and 258 participants in the nalmefene group

14. Secondary Outcome: Change in Clinical Status Using the CGI-I
Description: as for outcome 7
Time Frame: Week 52
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 95 | 258
units on a scale | 2.52 (0.10) | 2.26 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.029, Adjusted change from Baseline to Week 52; Mean Difference (Final Values) = -0.26, 95% CI [-0.50 to -0.03], Standard Error of Mean 0.12 — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Liver Function Test Gamma-glutamyl Transferase (GGT)
Description: GGT values
Time Frame: Week 52
Population: FAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 98 | 259
IU/L | 41.3 (76.2) | 32.0 (80.6)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.001, Adjusted values; Ratio to placebo = 0.78, 95% CI 2-sided [0.67 to 0.90] — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 98 participants in the placebo group and 259 participants in the nalmefene group

16. Secondary Outcome: Liver Function Test Alanine Aminotransferase (ALAT)
Description: ALAT values
Time Frame: Week 52
Population: FAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 97 | 259
IU/L | 27.8 (55.6) | 24.6 (58.5)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.037, Adjusted values; Ratio to placebo = 0.88, 95% CI 2-sided [0.79 to 0.99] — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 97 participants in the placebo group and 259 participants in the nalmefene group

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 52 weeks and a safety follow-up (visit/telephone call) scheduled for 4 weeks after completion of the study or after withdrawal from the study. Other Adverse Events: 52 weeks.
Arm/Group | Placebo | Nalmefene 18.06 mg
Serious Adverse Events (participants affected / at risk) | 8/164 | 35/501
Other Adverse Events (participants affected / at risk) | 57/164 | 273/501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=164) | Nalmefene 18.06 mg (N=501)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 9
Alcoholic hangover (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Anorexia nervosa (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arteritis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=164) | Nalmefene 18.06 mg (N=501)
Nausea (Gastrointestinal disorders) | 9 | 112
Vomiting (Gastrointestinal disorders) | 2 | 57
Fatigue (General disorders) | 3 | 27
Nasopharyngitis (Infections and infestations) | 19 | 54
Accidental overdose (Injury, poisoning and procedural complications) | 9 | 9
Fall (Injury, poisoning and procedural complications) | 11 | 5
Dizziness (Nervous system disorders) | 6 | 73
Headache (Nervous system disorders) | 13 | 61
Somnolence (Nervous system disorders) | 8 | 42
Insomnia (Psychiatric disorders) | 11 | 73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub publication. The investigators shall obtain Lundbeck's written approval before publishing any publication relating to nalmefene, the Study, the Protocol and/or the results recorded during the Study.